CLINICAL TRIAL: NCT00711581
Title: Evaluation of the Efficacy and Safety of the Endograb: A Laparoscopic Internal Retractor Device
Brief Title: Evaluation of Laparoscopic Internal Retractor Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endograb-HMO-CTIL
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2008-06

CONDITIONS: Cholelithiasis
Keywords: Cholecystectomy; Cholecystectomy, Laparoscopic; Laparoscopy
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Subjects will undergo a laparoscopic cholecystectomy. The gallbladder will be retracted using the Endograb retractor.
  Interventions: Device: Gallbladder retraction

INTERVENTIONS:
Device: Gallbladder retraction — The gallbladder will be retracted using the Endograb retractor
  Other Names: Endograb

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the Endograb system which is an internal laparoscopic retractor device. This retractor device is inserted into the abdominal cavity through one of the 5 mm trocars and obviates the need for a separate dedicated trocar for retraction. Therefore enables the reduction of the number of abdominal incisions in a laparoscopic operation.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic cholelithiasis
* Age 18-60
* ASA 1-2
* Able to sign an informed consent

Exclusion Criteria:

* ASA 3 or more
* Acute cholecystitis
* Choledocholithiasis
* Coagulation disorders
* Patients on blood thinners
* Use of Steroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Outcome will be either "success" or "failure". Success if the organ will be retracted adequately with the Endograb retractor. Failure if it will be necessary to add another trocar for inserting a retracting instrument. | 1 year

SECONDARY OUTCOMES:
No adverse effects related directly to the use of the Endograb retractor. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Mintz, MD, Principal Investigator — Hadassah Medical Organization; Ram Elazary, MD, Study Director — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Yoav Mintz, Jerusalem
  - Hadassah Medical Organization, Jerusalem